CLINICAL TRIAL: NCT05041634
Title: The Physical and Psychosocial Influences of an Exercise and Activity Program on People With Behavioral Diagnoses: A Cohort Study
Brief Title: Physical Activity for People With Behavioral Diagnoses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9088
Record Dates: First submitted 2021-09-03; First posted 2021-09-13 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Severe Mental Illness
Keywords: exercise, healthy habits, self-management
MeSH Terms: conditions — Mental Disorders; Motor Activity

STUDY DESIGN:
Intervention Model Description: pilot study of single group pre/post design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Group Pilot study pre/post (Experimental): One group of 8 participants receiving 14 week intervention
  Interventions: Behavioral: IHOPE

INTERVENTIONS:
Behavioral: IHOPE — Integrating Healthy Habits Optimized by Community Participation and Engagled Learning

SUMMARY:
Our aims are to 1) test that our intervention that can be measured with high fidelity. 2) determine the feasibility of the intervention including recruitment, procedures, measures, intervention acceptability and resources . 3)We will also test the outcomes of this 14-week fitness and wellness program based at a YMCA Healthy Living Center to gauge the effects of exercise and activity on patients with behavioral diagnoses including bipolar disorder, schizoaffective disorder, and schizophrenia. We also want to explore the influence of participating in such a program on the perceptions of mental illness among rehabilitation sciences students.

DETAILED DESCRIPTION:
Our aims are to 1) test that our intervention that can be measured with high fidelity. 2) determine the feasibility of the intervention including recruitment, procedures, measures, intervention acceptability and resources . 3)We will also test the outcomes of this 14-week fitness and wellness program based at a YMCA Healthy Living Center to gauge the effects of exercise and activity on patients with behavioral diagnoses including bipolar disorder, schizoaffective disorder, and schizophrenia. We also want to explore the influence of participating in such a program on the perceptions of mental illness among rehabilitation sciences students.

Our hypotheses are 1) that a fitness and activity program using physical activity, group discussion, and education delivered in a fitness facility will reduce anxiety and depression and strengthen hope, self-esteem, and improve overall quality of life; and 2) that student perceptions of mental illness will improve after participating in such a fitness and activity program.

Research Questions:

How does a program of exercise and activity influence the physical health of people with behavioural diagnoses as it relates to venous blood plasma measures of haemoglobin, cholesterol, lipids, insulin, glucose, triglycerides, high-density lipoproteins; height, weight, abdominal girth, blood pressure and heart rate; strength; and capacity for physical activity? How does a program of exercise and activity influence the psychosocial health of people with behavioural diagnoses as it relates to measures of hope, depression, anxiety, and self-esteem? How does a program of exercise and activity influence occupational performance and satisfaction of people with a behavioural diagnoses? How does a program of exercise and activity influence quality of life for people with a behavioral diagnoses ? How does participating in a program of exercise and activity influence the overall perceptions of people with behavioural diagnoses? What is the feasibility and fidelity of this 14-week intervention? How does being part of a program of exercise and activity for people with behavioural diagnoses influence perceptions of rehabilitation sciences students about mental illness?

EXPERIMENTAL DESIGN:

This follow up study involves a group of up to ten past participants recruited from patients being treated by the OU-Tulsa IMPACT Team. We will conduct interviews and baseline measures to compare to past progress. This study will serve to inform future cohorts for the original study protocol.

PROPOSED PROCEDURE:

Assessments include biophysical markers of health, self-reported psychosocial measures, and records of exercise and activity. Specifically, we will measure:

Cholesterol, lipids, and glucose/ A1C via blood specimens collected as a routine part of the patient's care Height and weight via stadiometer and digital scale, abdominal girth (the narrowest point between the xiphoid process and the navel) using a Gulick tape measure.

Blood pressure using a sphygmomanometer & heart rate by counting the pulse for 60 seconds using a digital timer Cardiovascular endurance via the three-minute step test Depression via the PHQ9 scale Anxiety using the Generalized Anxiety Disorder Test Interview/Focus Group Mental Illness Clinician Attitude Scale (MICA) This brief follow up study will assess participants who are one year out from the program or more. The study will take place in their residence and include the measures stated above and an interview. Researchers want to understand how the program is beneficial after one year and what can be improved to maintain benefits if any. Findings will be used to adjust the original protocol if needed to continue the original study. The assessments and interviews will be completed by researchers and occupational and physical therapy students under the supervision of their faculty. In addition, participants will be offered educational materials to help resume healthy habits.

ELIGIBILITY:
Inclusion Criteria:

All study participants will be over the age of 21 and will include women and likely some individuals who report minority status with a mental health diagnosis

Exclusion Criteria:

Under the age of 21 or who are not psychologically stable in the last month

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure | pre and post 14 week intervention
  self-rating goal tool
Coach Fidelity Log Sheet | first 8 weeks
  Coaches collected data for consistency of intervention
PHQ-9 | week1 and week 14
  self-rating depression screener
GAD | week1 and week 14
  Self-rated anxiety scale

OTHER OUTCOMES:
Blood Lipids | week1 and week 14
  hemoglobin, cholesterol, lipids, insulin, glucose, triglycerides, high-density lipoproteins;

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oklahoma Health Sciences Center, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No